CLINICAL TRIAL: NCT06467058
Title: Convergent Validity of the DABQ Questionnaire With the Actigraph as Reference Method to Assess 24-hour Movement Behaviors Among Adults
Brief Title: Convergent Validity of DABQ Questionnaire
Acronym: DABQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ONZ-2023-0384
Record Dates: First submitted 2024-02-26; First posted 2024-06-20 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Health Behavior
Keywords: convergent validity; Actigraph; Daily activity behavior questionnaire; 24-hour movement behaviors
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: convergent validity of a daily activity behavior questionnaire with the actigraph as reference among healthy adults
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adults (Other): In this study, participants will have one contact session with the researcher, which will be held either at Ghent University Hospital or at the participants' home. During this session, participants will be provided with an accelerometer device and two questionnaires (to be filled in after wearing the Actigraph), namely the Daily Activity Behavior Questionnaire (DABQ) and general information questionnaire.
  The participants will receive an Actigraph wGT3X+BT accelerometer which will be worn for seven consecutive days. Instructions will be given on how to wear the accelerometer (e.g. during the day at the hip and during the night at the wrist). At the end of this week, the participants will fill in both questionnaires. After wearing the accelerometer for seven consecutive days and filling in both questionnaires, the researcher will visit the participants to collect the devices, or the participants will send them back by postal package.
  Interventions: Device: DABQ questionnaire versus Actigraph as reference method

INTERVENTIONS:
Device: DABQ questionnaire versus Actigraph as reference method — In this study, participants will have one contact session with the researcher, which will be held either at Ghent University Hospital or at the participants' home. During this session, participants will be provided with an accelerometer device and two questionnaires (to be filled in after wearing the Actigraph), namely the Daily Activity Behavior Questionnaire (DABQ) and general information questionnaire.
  The participants will receive an Actigraph wGT3X+BT accelerometer which will be worn for seven consecutive days. Instructions will be given on how to wear the accelerometer (e.g. during the day at the hip and during the night at the wrist). At the end of this week, the participants will fill in both questionnaires. After wearing the accelerometer for seven consecutive days and filling in both questionnaires, the researcher will visit the participants to collect the devices, or the participants will send them back by postal package.

SUMMARY:
Time-use epidemiology is a rapidly growing research area that aims to understand how individuals allocate their time to various activities throughout the day. Accurate assessment of daily activity behaviors, such as sleep, sedentary behavior (SB), light physical activity (LPA), and moderate to vigorous physical activity (MVPA), is crucial for studying the associations between activity patterns and health outcomes. To gather this information, researchers often rely on self-report questionnaires and objective measures, such as accelerometers, to provide a comprehensive understanding of individuals' activity levels.

Recently, a validated questionnaire known as the Daily Activity Behavior Questionnaire (DABQ) has been developed. In a study comparing DABQ estimates with the activPAL4 accelerometer (as the reference method), good results regarding absolute agreement and consistency were obtained for sleep duration (ICC 0.6), while the absolute agreement and consistency for SB, LPA, and MVPA estimates was lower (ICC ranging from 0.22-0.47).

It should be noted that this study acknowledges the limitation of not treating the data as compositional data. Compositional data analysis accounts for the relative distribution of different activities and avoids the assumption of independence between behaviors. Additionally, the activPAL4 accelerometer used as the reference method in the study had its own strengths and weaknesses when compared to other objective measures, such as the Actigraph. Where ActivPAL4 is more used to differentiate between sitting and standing, Actigraph is able to better classify activity intensities. Moreover, as recommended in different research, I use the Actigraph in my PhD to objectively asses 24-hour movement behaviors.

Given these considerations, the aim of this study is to validate the DABQ against the Actigraph as the reference method. Furthermore, this study aims to analyze the data as compositional data, which would provide a more comprehensive understanding of the interrelatedness of behaviors. The hypothesis is that there will be moderate convergent validity between the DABQ and Actigraph, allowing for accurate assessment of sleep duration, SB, LPA, and MVPA. By establishing the validity of the DABQ and considering the data as compositional, researchers can utilize this questionnaire in time-use epidemiology studies, which could be seen as an easy to use and cost-effective measurement method.

ELIGIBILITY:
Inclusion Criteria:

- Adults between 18 and 65 years old

Exclusion Criteria:

* Physical (e.g. amputations, paralysis, recovering from stroke, osteoarthritis conditions that obstruct daily functioning
* Cognitive (e.g. dementia, psychological disorders) conditions that obstruct daily functioning
* Major medical (e.g. Chronic respiratory diseases, heart failure, cardiovascular diseases) conditions that obstruct daily functioning

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-09-30 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Total 24-hour movement behaviors collected by the Actigraph GT3X+BT | Through study completion, an average of 2 weeks
  The Actigraph GT3X+BT will objectively collect time spent in sleep, sedentary behavior and physical activity. This device will be worn be the participants during 7 consecutive days (at night at their non-dominant wrist and during the day at their right hip).
Total 24-hour movement behaviors collected by the Daily Activity Behavior Questionnaire (DABQ) | Through study completion, an average of 2 weeks
  This questionnaire will subjectively collect time spent in sleep, sedentary behavior and physical activity. This questionnaire will be filled in at the end of the 7 days wearing the Actigraph mentioned in outcome 1.
Convergent validity between time spent in 24-hour movement behaviors collected by the Actigraph GT3X+BT and DABQ | Through study completion, an average of 2 weeks
  Intraclass correlation coefficient (95% confidence intervals) and pearson/spearman correlation will be used to measure the convergent validity and intermeasurement reliability. This method allows the comparison between self-reported use of time and the device measured use of time for each behavior separately.

SECONDARY OUTCOMES:
Participant characteristics "sex" potentially explaining biases in reporting 24-hour movement behaviors. | Through study completion, an average of 2 weeks
  Interaction effects between difference in measurement (Actigraph versus DABQ) and participant characteristics are explored to better interpret discrepancies between questionnaire- and accelerometer-assessed physical activity, ensuring more reliable and generalizable findings.
Participant characteristics "age" potentially explaining biases in reporting 24-hour movement behaviors. | Through study completion, an average of 2 weeks
  Interaction effects between difference in measurement (Actigraph versus DABQ) and participant characteristics are explored to better interpret discrepancies between questionnaire- and accelerometer-assessed physical activity, ensuring more reliable and generalizable findings.
Participant characteristics "body mass index" potentially explaining biases in reporting 24-hour movement behaviors. | Through study completion, an average of 2 weeks
  Interaction effects between difference in measurement (Actigraph versus DABQ) and participant characteristics are explored to better interpret discrepancies between questionnaire- and accelerometer-assessed physical activity, ensuring more reliable and generalizable findings.
Participant characteristics "family situation" potentially explaining biases in reporting 24-hour movement behaviors. | Through study completion, an average of 2 weeks
  Interaction effects between difference in measurement (Actigraph versus DABQ) and participant characteristics are explored to better interpret discrepancies between questionnaire- and accelerometer-assessed physical activity, ensuring more reliable and generalizable findings.
Participant characteristics "children" potentially explaining biases in reporting 24-hour movement behaviors. | Through study completion, an average of 2 weeks
  Interaction effects between difference in measurement (Actigraph versus DABQ) and participant characteristics are explored to better interpret discrepancies between questionnaire- and accelerometer-assessed physical activity, ensuring more reliable and generalizable findings.
Participant characteristics "educational level" potentially explaining biases in reporting 24-hour movement behaviors. | Through study completion, an average of 2 weeks
  Interaction effects between difference in measurement (Actigraph versus DABQ) and participant characteristics are explored to better interpret discrepancies between questionnaire- and accelerometer-assessed physical activity, ensuring more reliable and generalizable findings.
Participant characteristics "sedentary job" potentially explaining biases in reporting 24-hour movement behaviors. | Through study completion, an average of 2 weeks
  Interaction effects between difference in measurement (Actigraph versus DABQ) and participant characteristics are explored to better interpret discrepancies between questionnaire- and accelerometer-assessed physical activity, ensuring more reliable and generalizable findings.
Participant characteristics "net family income" potentially explaining biases in reporting 24-hour movement behaviors. | Through study completion, an average of 2 weeks
  Interaction effects between difference in measurement (Actigraph versus DABQ) and participant characteristics are explored to better interpret discrepancies between questionnaire- and accelerometer-assessed physical activity, ensuring more reliable and generalizable findings.
Participant characteristics "smoking status" potentially explaining biases in reporting 24-hour movement behaviors. | Through study completion, an average of 2 weeks
  Interaction effects between difference in measurement (Actigraph versus DABQ) and participant characteristics are explored to better interpret discrepancies between questionnaire- and accelerometer-assessed physical activity, ensuring more reliable and generalizable findings.
Participant characteristics "feasibility of wearing the Actigraph" potentially explaining biases in reporting 24-hour movement behaviors. | Through study completion, an average of 2 weeks
  Interaction effects between difference in measurement (Actigraph versus DABQ) and participant characteristics are explored to better interpret discrepancies between questionnaire- and accelerometer-assessed physical activity, ensuring more reliable and generalizable findings.
Participant characteristics "annoying to wear the Actigraph" potentially explaining biases in reporting 24-hour movement behaviors. | Through study completion, an average of 2 weeks
  Interaction effects between difference in measurement (Actigraph versus DABQ) and participant characteristics are explored to better interpret discrepancies between questionnaire- and accelerometer-assessed physical activity, ensuring more reliable and generalizable findings.
Participant characteristics "consistency of wearing the Actigraph" potentially explaining biases in reporting 24-hour movement behaviors. | Through study completion, an average of 2 weeks
  Interaction effects between difference in measurement (Actigraph versus DABQ) and participant characteristics are explored to better interpret discrepancies between questionnaire- and accelerometer-assessed physical activity, ensuring more reliable and generalizable findings.

CONTACTS AND LOCATIONS:
Overall Officials: Marieke De Craemer, Principal Investigator — University Ghent
Locations (1):
- Ghent university Hospital, Ghent, Belgium